CLINICAL TRIAL: NCT04065581
Title: Randomized, Non-blinded Crossover Study to Establish the Bioequivalence Between Fixed Dose Combination (FDC) and the Loose Combination of Acarbose and Metformin Following Single Oral Dosing in Chinese Healthy Adult Male and Female Subjects
Brief Title: Bioequivalence Study for Acarbose/Metformin FDC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19843
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A-washout-treatment B (Experimental): Subject will receive a single oral dose of acarbose/metformin FDC (Treatment A, 50 mg acarbose/500 mg metformin) in period 1, followed by a single oral dose of 50mg acarbose and 500mg metformin as loose combination (Treatment B) in period 2. Washout interval between 2 treatment periods was at least 7 days.
  Interventions: Drug: Acarbose/Metformin FDC(BAY81-9783); Drug: Glucobay; Drug: Glucophage
- Treatment B-washout-treatment A (Experimental): Subject will receive a single oral dose of 50 mg acarbose and 500 mg metformin as loose combination (Treatment B) in period 1, followed by a single oral dose of acarbose/metformin FDC (Treatment A, 50mg acarbose/500 mg metformin) in period 2. Washout interval between 2 treatment periods was at least 7 days.
  Interventions: Drug: Acarbose/Metformin FDC(BAY81-9783); Drug: Glucobay; Drug: Glucophage

INTERVENTIONS:
Drug: Acarbose/Metformin FDC(BAY81-9783) — Single dose: 50 mg acarbose/500 mg metformin tablet, oral
Drug: Glucobay — Single dose: 50 mg tablet, oral
Drug: Glucophage — Single dose: 500 mg tablet, oral

SUMMARY:
The purpose of this study is to establish the bioequivalence (i.e. similar pharmacokinetics and pharmacodynamics characteristics) between acarbose/metformin FDC (50 mg/500 mg) and loose combination of acarbose (50 mg) and metformin (500 mg)

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male or non-pregnant, non-lactating female subject, age ≥ 18 years at the first screening examination / visit.
* Body Mass Index (BMI): ≥ 19 to <28 kg / m*2 , with body weight ≥ 50 kg.
* Results of HbA1c value are within the normal range (4.0-6.0%, inclusive).
* Plasma glucose after 75g oral glucose loading show:

  * FPG (Fast Plasma Glucose) < 6.1 mmol / dL.
  * 2-h PG (Plasma Glucose 2 hours after glucose loading) < 7.8 mmol/dL
* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time phase between signing of the informed consent form and the last visit. The acceptable methods of contraception available to men include, for example (e.g.) condoms with or without a spermicidal agent; the acceptable methods of contraception available to women include e.g. (a) diaphragm or cervical cap with spermicide; (b) intra-uterine device; (c) hormone-based contraception (only for the female partners of male subjects) One method has to be used by the man and one method by the female partner. No need to use two methods at the same time if subject or his female partner has been surgically sterilized ,
* Subjects who are able to understand and follow instructions and who are able to participate in the study for the entire period
* Subjects must give their written informed consent to participate in the study after receiving adequate previous information and prior to any study specific procedures

Exclusion Criteria:

* Screening test results likely to show inappropriateness for participation in this study:

  * Any clinically relevant abnormality identified on the screening medical examination
  * Systolic blood pressure < 90 or ≥ 140 mmHg (after at least 5 min in supine position)
  * Diastolic blood pressure < 60 or ≥ 90 mmHg (after at least 5 min in supine position)
  * Pulse rate < 50 or > 100 beats/min (after at least 5 min in supine position)
  * Clinically relevant findings in the electrocardiogram (ECG) such as a second- or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QTcB-interval over 450 msec
  * Positive results for hepatitis B virus surface antigen (hepatitis B surface antigene (HBsAg)), hepatitis C virus antibodies (anti-HCV) and human immune deficiency virus antibodies (human immunodeficiency virus antibodies (anti-HIV)) and treponema pallidum specific antibody.
  * Positive urine drug screening
  * Hemoglobin level lower than Lower limit of normal value
  * Clinical laboratory results evaluated by the investigators to be clinically abnormal values
* A history of relevant diseases of internal organs (diabetes mellitus, Ileus, Ileus-like symptoms, diseases that may significantly jeopardize body systems, such as malabsorption or maldigestion from gastrointestinal tract, liver cirrhosis, renal dysfunction, congestive heart failure, ischemic heart disease, malignant neoplasm), of the central nervous system (e.g. epilepsy), or other organs which are likely to show inappropriateness for participation in this study
* States which may deteriorate as a result of increased gas formation in the intestine (e.g. Roemheld's syndrome, major hernias, intestinal obstructions, and intestinal ulcers).
* Acute conditions with the potential to alter renal function such as: dehydration, severe infection, shock.
* Any type of acute metabolic acidosis.
* Family history of diabetes (within the second degree of relationship)
* Known drug hypersensitivity or idiosyncrasy
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Special diets or known hypersensitivity preventing the subjects from eating the standard meals during the study.
* Habitual medication including Chinese herbal drugs within 3 months before the screening
* Participation in another clinical trial within 3 months before the screening examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
RatioCmax (serum glucose) | Treatment period 1 and 2, Day-1 and Day 1: 10 minutes, 25 minutes, 40 minutes, 55 minutes, 1 hour 10 minutes, 1 hour 40 minutes, 2 hours 10 minutes, 3 hours 10 minutes, 4 hours 10 minutes
  RatioCmax=Cmax,day1/ Cmax,day-1 Cmax,day-1: Maximum serum glucose after 75g sucrose loading on Day -1 Cmax,day1: Maximum serum glucose after 75g sucrose loading and single dose administration of study drug on Day 1
RatioAUC(0-4) (serum glucose) | Treatment period 1 and 2, Day-1 and Day 1: 10 minutes, 25 minutes, 40 minutes, 55 minutes, 1 hour 10 minutes, 1 hour 40 minutes, 2 hours 10 minutes, 3 hours 10 minutes, 4 hours 10 minutes
  RatioAUC(0-4)=AUC(0-4),day1/AUC(0-4),day-1 AUC (0-4),day1: AUC of serum glucose from time 0 to 4 hours on Day 1 AUC(0-4),day-1: AUC of serum glucose from time 0 to 4 hours on Day -1
Cmax (plasma metformin) | Treatment period 1 and 2: Pre-dose, 0.5 hour, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 24 hours
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration / maximum drug concentration in plasma after single dose administration
AUC (0-tlast) (plasma metformin) | Treatment period 1 and 2: Pre-dose, 0.5 hour, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 24 hours
  AUC (0-tlast): AUC from time 0 to the last data point > LLOQ (lower limit of quantification)
AUC (plasma metformin) | Treatment period 1 and 2: Pre-dose, 0.5 hour, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 24 hours
  AUC: Area under the concentration vs. time curve from zero to infinity after single (first) dose

SECONDARY OUTCOMES:
Frequency of TEAE (treatment-emergent adverse event） | Approximate 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal